CLINICAL TRIAL: NCT06721143
Title: A Double-blinded, Randomized, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of AION-301 Administered by Intravenous Infusion for the Treatment of Participants with Stage 3 Chronic Kidney Disease
Brief Title: A Study to Investigate the Safety, Tolerability, and Preliminary Efficacy with AION-301 Administered by Intravenous Infusion Compared with Placebo Administered by Intravenous Infusion Investigational Intervention in Participants Aged 35 to 75 Years of Age with Chronic Kidney Disease (CKD)
Acronym: UC-MSC-CKD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AION Healthspan, Inc. (Industry)
Collaborators: George Clinical (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AION-301-CKD-2024
Record Dates: First submitted 2024-11-07; First posted 2024-12-06 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Disease Stage 3
Keywords: CKD; AION-301; Stage 3 CKD; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Active Comparator): AION-301
  Interventions: Biological: AION-301
- Group II (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: AION-301 — AION-301 Infusion
  Arms: Group I
Drug: Placebo — Placebo Infusion
  Arms: Group II

SUMMARY:
The goal of this clinical trial is to learn about the safety (good or bad) of giving two AION-301 intravenous (IV) infusions, in adults with Stage 3 Chronic Kidney Disease (CKD). It will also help to learn if AION-301 reduces the symptoms of CKD and/or progression. The main questions it aims to answer are:

* Do participants have medical problems (adverse events) after receiving two infusions of AION-301?
* Do participants feel better (have reduced and/or delayed CKD symptoms)?
* To learn about how AION-301 works in participants with CKD?

Researchers will compare AION-301 to a placebo (a look-alike substance that contains no drug) to see if AION-301 works to treat Stage 3 CKD.

Participants will:

* Receive two infusions of AION-301 or placebo on two separate days (Day 0 and Day 4).
* Receive oral vitamins at the clinic and to take at home for 90 days.
* Visit the clinic for a minimum of 9 times, over 6 months for checkups and tests, but could be up to 12 times, over 24 months for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Patient is able to communicate well with the investigator, is capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol, understands all requirements of the study, and understands and signs the written ICF before any study-specific procedure.
* Willing and able to comply with the scheduled visits and treatment plan.
* Either biological sex
* Participant must be 35 to 75 years of age inclusive, at the time of signing the informed consent.
* Diagnosis of CKD stage 3, G3 (a and b): persistent eGFR between 30 and 59 mL/min/1.73 m² (at least 2 measures within that range in the preceding 3 months, including the one at screening visit), and persistent increased Albuminuria (at least 2 measures within 3 months, including 1 before screening and 1 at screening (criterion for increased Albuminuria at screening: ≥2 out of 3 repeat daily early morning samples at screening) (UACR ≥ 200 mg/g and < than 5000 mg/g)
* Treatment with maximum labelled or tolerated dose of a renin-angiotensin-aldosterone system (RAAS) blocking agent including an angiotensin converting enzyme (ACE) inhibitor or an angiotensin II receptor blocker (ARB), and SGLT2 inhibitors (SGLT2i) unless such treatment is contraindicated or not tolerated*. Treatment dose must be stable for at least 3 months prior to the date of the screening. If a patient is on treatment with GLP-1 receptor agonist, he/she should be on a stable dose for at least 3 months before screening.

  *Participants who are documented to be unable to take ACE inhibitors or ARBs or SGLT2i will be allowed to participate.
* Female subjects must not be breastfeeding and must have no intention to become pregnant during the study, and she will be required to use at least two FDA approved birth control during the study. The FDA-approved and cleared methods for birth control are listed below:

  * Permanent Sterilization
  * Long-Acting Reversible Contraceptives (LARC)
  * Contraceptive Injection
  * Short-Acting Hormonal Methods
  * Barrier Methods
  * Emergency Contraception
* Any male subject must agree to use contraceptives and not donate sperm during the study.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Prior transplant of any organ (including BM and stem cell transplant) or kidney transplant scheduled in the next 6 months.
* Proteinuria>5000 and or serum Albumin< 2.5 g/dl.
* Acute coronary syndrome, stroke or TIA or hospitalization for heart failure in previous 12 weeks or poorly controlled hypertension (≥160/100 mmHg at screening visit) or SBP<90 at screening visit.
* History of malignancy (except successfully treated squamous and basal cells skin carcinoma) within 5 years of screening.
* History of atrial fibrillation (AF, AFib).
* CKD due to genetic disorder.
* History of systemic Autoimmune diseases like T1D, SLE or CKD caused by any autoimmune kidney disease.
* Acute Kidney Injury (AKI) defined as increase in serum creatinine ≥1.5 times baseline in the previous 3 months or by presence of acute tubular injury in kidney biopsy in the previous 3 months.
* Dialysis for acute renal failure within 12 weeks of screening visit.
* Rapidly progressive kidney disease (eGFR reduction ≥ 30% over the last three months)
* HbA1c ≥ 8.5%.
* BMI ≥35 kg/m2.
* Disorder of coagulation (including any history of thrombotic or thromboembolic disease) and/or long-term anti-coagulant therapy
* History of Deep Vein Thrombosis (DVT)
* History of Acute Pulmonary Embolism
* History of solitary kidney.
* On medications such as immunosuppressant, monoclonal antibodies, anabolic steroids, at the time of screening or in the previous 6 months and/or illicit drugs.
* History of alcohol abuse or cigarette smoking in the previous 6 months.
* Pregnancy or breast feeding at the time of screening, or with intention to become pregnant or breast-feeding during the course of the study, including the follow-up period.
* History of liver disease, ALT and AST ≥3 x ULN, positive serology for Hepatitis B or Hepatitis C, HIV.
* A significant medical history or abnormality at the physical exam that, in the judgment of the principal investigator, may interfere with the study.
* Presence of any active infection, including COVID 19
* Any clinically significant pulmonary disease
* History of hypersensitivity to study drug and/or any of its excipients.
* Close affiliation with the investigational site; for example, a close relative of the investigator, dependent person (for example employee or student of the investigational site).
* Panel Reactive Antibodies (PRA) >0% (positive)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Treated Participants Experiencing Grade 3 or Above Adverse Events As Assessed by CTCAE V5.0 | From baseline through day 90
  The primary analysis will be to test safety and tolerability AION-301 DP treatment in patients with CKD as assessed by the proportion of patients experiencing adverse events grade 3 or above (based on CTCAE version 5) by day 90 following treatment in comparison with Placebo group. This will be conducted by the unblinded trial biostatistician using standard two sample tests of proportions such as chi-squared tests or Fisher's exact tests.

SECONDARY OUTCOMES:
To assess the potential evidence of efficacy in participants by | From Baseline for up to 2 years
  The differences between groups in the proportion of patients with reduced proteinuria.
To assess the potential evidence of efficacy in participants by | From Baseline for up to 2 years
  Evaluations of effects and persistence of effects by measuring Urinary Albumin-to-Creatinine Ratio (UACR), Urinary Protein-to-Creatinine Ratio (UPCR), and estimated Glomerular Filtration Rate (eGFR).
To assess the potential evidence of efficacy in participants by | From Baseline for up to 2 years
  The impact of treatment on Quality of Life with the KDQOL-36 questionnaire.
KidneyIntelX Risk Profile | From baseline through 6 months
  Changes in KidneyIntelX risk levels

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami, Leonard M. Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided